CLINICAL TRIAL: NCT00836251
Title: Effects of Antipsychotic Medications on Energy Intake and Expenditure
Acronym: DLW
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 06-0246
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Weight Gain
Keywords: energy expenditure; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- H218O and 2H2O: schizophrenia
  Interventions: Dietary Supplement: H218O and 2H2O, administered as a mixed cocktail

INTERVENTIONS:
Dietary Supplement: H218O and 2H2O, administered as a mixed cocktail — 0.195 g of H218O and 0.117 g of 2H2O per kg of estimated total body water (TBW), administered as a mixed cocktail

SUMMARY:
Aim 1: To evaluate the effect of antipsychotic treatment group on Activity Energy Expenditure. The project hypothesizes that subjects treated with olanzapine will demonstrate a greater decrease in AEE over time than subjects treated with ziprasidone, due at least in part to sedating effects of olanzapine.

Aim 2: To evaluate the effect of antipsychotic treatment group on Energy Intake. The project hypothesizes that subjects treated with olanzapine will demonstrate a greater increase in EI over time than subjects treated with ziprasidone, based on higher histamine type 1 (H1) receptor affinity of olanzapine and the relationship between H1 affinity and hunger and/or satiety.

DETAILED DESCRIPTION:
The overall purpose of this research is to determine how two commonly prescribed antipsychotic medications, olanzapine (Zyprexa) and ziprasidone (Geodon), affect weight gain through increasing appetite and/or through increasing sedation that results in decreased activity.

Undesirable changes in body weight, blood sugar control, type 2 diabetes, and blood lipids occur more commonly in people who have schizophrenia than in people without psychiatric conditions. Although differences in glucose regulation were first reported in schizophrenia before the use of antipsychotic medications, antipsychotic treatment may contribute to these problems, though just how this happens is not understood. This study proposes to use a doubly-labeled water (DLW) method to measure the degree to which weight gain (fat mass) is due to increased appetite, decreased physical activity from being tired and sleepy, or some combination of both. Doubly-labeled water contains stable isotopes (non-radioactive forms) of the hydrogen and oxygen that make up all water, isotopes that will be slowly passed out through the urine after participants drink DLW. The number of hydrogen and oxygen isotopes found in the urine samples will tell us how many calories the participant's body has been using.

The DLW method has been used in people with obesity and other types of medical problems. It's recognized as the most accurate measure of the number of calories burned throughout a typical day, and how many calories are taken in from food and drink. By measuring these factors in people who take antipsychotic medications, doctors will gain a better understanding of the effects of antipsychotic medications on body weight and fat mass. This could lead to the development of better ways to prevent or treat weight gain or diabetes in patients who take antipsychotic medications.

ELIGIBILITY:
Inclusion Criteria:

* non-diabetic
* schizophrenic or schizoaffective
* currently prescribed olanzapine or ziprasidone
* 18-80 y.o.

Exclusion Criteria:

* <18 or >80 years of age
* diabetic
* not schizophrenic or schizoaffective
* not currently prescribed olanzapine or ziprasidone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females, ages 18-80, diagnosed with schizophrenia or schizoaffective disorder
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
treatment-induced changes in Total Energy Expenditure (TEE), Activity Energy Expenditure (AEE), and Energy Intake (EI) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John W Newcomer, MD, Principal Investigator — Florida Atlantic University; Ginger Nicol, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States